CLINICAL TRIAL: NCT03807427
Title: Using Adapted Dialectical Behavior Skills as Mental Health Prevention in Post-Earthquake Nepal: READY-Nepal Protocol for a Pilot Feasibility and Acceptability Trial
Brief Title: Regulating Emotions Through Adapted Dialectical Behavior Skills for Youth (READY-Nepal)
Acronym: READY-Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandon A Kohrt, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Brandon A Kohrt, MD, PhD, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00071881
Record Dates: First submitted 2019-01-03; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Mental Disorders
Keywords: Adolescents; Mental Health; Prevention; Emotion Regulation; Global Mental Health
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- READY-Nepal (Experimental): Skills groups based on dialectical behavior therapy principles delivered over 10-12 weeks in a classroom format.
  Interventions: Behavioral: READY-Nepal
- Waitlist Control (No Intervention): Adolescent participants assigned to the control condition will be placed on a waitlist for future enrollment in READY-Nepal. After primary data collection has ceased, those assigned to the control arm will receive the identical READY-Nepal intervention delivered in the experimental condition.

INTERVENTIONS:
Behavioral: READY-Nepal — Regulating Emotions through Adapted Dialectical behavior skills for Youth in Nepal (READY-Nepal) is a brief (10-session), emotion-focused intervention targeting prevention and reduction of trans diagnostic problems related to emotion regulation. The culturally adapted program is divided into 5 modules, and includes both didactic and experiential instruction in skills related to mindfulness, stress tolerance, emotional awareness and regulation, validation of self and others, and mastery of interpersonal relationships.
  Other Names: Adolescent Emotion Dysregulation Prevention Intervention
  Arms: READY-Nepal

SUMMARY:
Published research on the development of mental health symptomatology among adolescents has expanded in recent years and indicates the presence of a growing public health concern. The 2015 earthquakes in Nepal are a risk factor for increased psychological distress across all age groups. Prior studies have also demonstrated high chronic risk of suicidal thoughts and behaviors (STBs) among adolescents in Nepal and throughout South Asia. Despite the need for mental health promotion interventions in Nepal, there is a lack of psychological treatments for suicide prevention that have been rigorously evaluated in Nepal. To address this gap, a trans diagnostic, emotion -focused mental health promotion intervention (Regulating Emotions through Adapted Dialectical behavior skills for Youth in Nepal; READY-Nepal) was developed for delivery in school-based settings. A pilot quasi-experimental trial utilizing a wait-list control group will be used to evaluate the feasibility and acceptability of the intervention in a cohort of school -going adolescents in the Kathmandu Valley. Qualitative methodology will be used to augment quantitative findings via exploration of gender differences in perception and uptake of the program, program feasibility and acceptability, as well as changes in coping skills and explanatory models of stress between baseline and follow- up. This pilot study will aid in modifying the intervention to inform the development of a larger, adequately powered cluster randomized trial (CRT) of READY-Nepal.

DETAILED DESCRIPTION:
SETTING: The study will be conducted in school settings in earthquake -affected areas throughout the Kathmandu Valley. Due to an aggregation of factors including political and environmental trauma, these areas are at high risk for the development and continuation of mental health problems.

STUDY DESIGN: Regulating Emotions through Adapted Dialectical behavior skills for Youth in Nepal (READY-Nepal) is a pilot quasi-experimental trial. All students between the ages of 13 to-17 enrolled in a secondary school in one of two earthquake -affected districts in the Kathmandu Valley will be eligible for participation. After enrollment, classes will be assigned to either READY-Nepal or a wait-list control condition. Groups will be gender-stratified due to concerns around stigma and confidentiality found in similar trials in Nepal and other low- and middle-income countries (LMIC). Because of the higher potential for contamination effects (i.e., transmission of skills or related intervention content) at the individual level, whole classroom sections will either be assigned to the experimental or waitlist conditions. Because of the pilot nature of this preliminary feasibility and acceptability trial, the sample size will not be powered for inference testing. Results from this pilot study will be used to identify parameters necessary for an appropriately powered cluster- randomized trial (CRT) of the intervention.

INTERVENTIONS: READY-Nepal is a 10 -session, classroom- based skills training program designed to promote positive mental health in addition to supporting resilient responses in trauma- exposed adolescents. The modularized, emotion-focused intervention was informed by principles of Dialectical Behavior Therapy (DBT) and was designed to augment and generalize Nepali adolescents' emotion regulation abilities during current or future stressful circumstances. READY-Nepal is divided into 5 components, and includes both didactic and experiential instruction in skills related to mindfulness, stress tolerance, emotional awareness and regulation, validation of self and others, and mastery of interpersonal relationships. The program was designed with a flexible delivery format in mind, in order to increase its dissemination potential in LMIC like Nepal. The program was developed from a prior, more intensive version of the intervention that was culturally adapted and piloted with self -destructive women in rural Nepal. READY-Nepal will be delivered by local Nepali clinical counselors trained by a US psychiatrist and clinical psychology doctoral student with comprehensive DBT training. Program facilitators will participate in weekly ongoing supervision with the original program developers.

PARTICIPANTS: School- going adolescents (ages 13- to 17) residing in earthquake-exposed areas in Kathmandu Valley are the intended direct beneficiaries of READY-Nepal. For this feasibility and acceptability pilot, additional qualitative component participants will include school teachers and primary caregivers of a subset of participating adolescents.

PLANNED ANALYSES Statistical analyses: Primary and secondary outcomes of interest will be summarized descriptively and visually over time for both study arms. Total and validated domain- specific scores will be evaluated for each instrument. Outcomes will be analyzed for within -group factor and intervention as a between- group factor. Preliminary estimates of within- and between -group variances and the intra-class correlation coefficient (ICC) of participant outcomes will be estimated and used to determine sample size calculations for a future, adequately powered cluster -randomized trial.

Qualitative analyses: qualitative research methodology and commercial software (NVIVO 9) will be used to analyze data from focus group discussions and in depth interviews. This method will consist of (1) reading each transcript multiple times for content, then (2) open coding transcripts for data on key themes surrounding the concepts of intervention effectiveness, stress -based explanatory models, and gender- moderated skills uptake. These coding segments will be combined into axial coding categories. The same, iterative process will continue for the remaining transcripts until a final set of emergent themes is presented. Checks for inter-rater reliability using kappa coefficients will also be performed.

ETHICS & RESEARCH GOVERNANCE Consent: Permission for conducting the program in each school will be obtained from school principals. For adolescent participants, research assistants will obtain participant as well as primary caregiver consent. Research assistants will also consent all adult participants participating in qualitative evaluation. All participants will have the opportunity to ask questions related to the process or to study elements. Subjects can also request a virtual or in person meeting with either the researchers or the principal investigator if additional questions arise at any point during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Students in the intervention and control arms are eligible for enrollment if they are between the ages of 13-17. Recruitment will attempt to balance gender and age distribution. All adolescent participants will need to be formally enrolled in a participating school.
2. Adults participating in qualitative evaluation must be fluent in Nepali. Parents are eligible if their child is an active participant in the program, and teachers are eligible if their students are current participants.

Exclusion Criteria:

1. There are no additional exclusion criteria.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Emotion Regulation | 1-week post-intervention
  Adolescent emotion regulation will be assessed using the Difficulties in Emotion Regulation Scale (DERS). The DERS has been transculturally adapted in Nepal for use with this population.

SECONDARY OUTCOMES:
Change in Anxiety | 1-week post-intervention
  Adolescent anxiety is assessed with the Nepali version of the Beck Anxiety Inventory (BAI). This instrument has been clinically and culturally validated for use in Nepal.
Change in Individual Coping | 1-week post-intervention
  Generalization of coping skills use will be assessed through the Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL). In Nepal, the instrument has been transculturally adapted and tested with a sample of suicidal and self-harming women.
Change in Depression | 1-week post-intervention
  Depression symptoms will be measured using a subset of items from the Nepali version of the Primary Care Depression Screening (PCDS). The PCDS has been clinically and culturally validated for use in Nepal.
Change in Post-Traumatic Stress | 1-week post-intervention
  Symptoms of post-traumatic stress will be assessed using a subset of items from the Nepali version of the Child PTSD Symptom Scale (CPSS). The CPSS has been clinically and culturally validated for use in Nepal.
Change in Self-Validation | 1-week post-intervention
  Adolescent self-validating behaviors will be assessed using the Self-Validating & Invalidating Questionnaire (SVSI-Q). This instrument has been culturally adapted for use in Nepal.
Change in Adolescent Functioning | 1-week post-intervention
  Adolescent functional impairment will be measured using the Nepali version of the Child Functioning Impairment Scale (CFI). The CFI has been clinically and culturally validated for use in Nepal.
Change in Resilience | 1-week post-intervention
  Adolescent resilience will be measured using items adapted from the Resilience Scale. This adapted scale has been clinically and culturally validated in Nepal.
Change in Implicit Self-Esteem | 1-week post-intervention
  Implicit self-esteem will be assessed using a computer-based Implicit Association Test (IAT). The Rosenberg Self-Esteem Scale (RSES) will be used as the standardized comparison tool for the IAT.
Change in Suicidal and Self-Harming Behaviors | 1-week post-intervention
  Suicidal ideation, suicide, and non-suicidal self-injury (NSSI) will be assessed via a 7-item scale including Depression Self-Rating Scale (DSRS) item #10, in addition to daily diary cards completed by participating adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Kohrt, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Transcultural Psychosocial Organization, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available upon request after publication of primary outcome results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be shared within 60 months of trial completion
Access Criteria: Contact principal investigator

REFERENCES:
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Bridge JA, Goldstein TR, Brent DA. Adolescent suicide and suicidal behavior. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):372-94. doi: 10.1111/j.1469-7610.2006.01615.x. PMID 16492264
- [Background] Corbin J, Strauss A. Basics of qualitative research: Techniques and procedures for developing grounded theory. Sage publications; 2014 Nov 25.
- [Background] Cousins S. Nepal's silent epidemic of suicide. Lancet. 2016 Jan 2;387(10013):16-7. doi: 10.1016/S0140-6736(15)01352-5. No abstract available. PMID 26766336
- [Background] Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of psychopathology and behavioral assessment. 2004 Mar 1;26(1):41-54.
- [Background] Kerres Malecki C, Kilpatrick Demary M. Measuring perceived social support: Development of the child and adolescent social support scale (CASSS). Psychology in the Schools. 2002 Jan 1;39(1):1-8.
- [Background] Kohrt BA, Jordans MJ, Tol WA, Luitel NP, Maharjan SM, Upadhaya N. Validation of cross-cultural child mental health and psychosocial research instruments: adapting the Depression Self-Rating Scale and Child PTSD Symptom Scale in Nepal. BMC Psychiatry. 2011 Aug 4;11(1):127. doi: 10.1186/1471-244X-11-127. PMID 21816045
- [Background] Kohrt BA, Jordans MJ, Tol WA, Speckman RA, Maharjan SM, Worthman CM, Komproe IH. Comparison of mental health between former child soldiers and children never conscripted by armed groups in Nepal. JAMA. 2008 Aug 13;300(6):691-702. doi: 10.1001/jama.300.6.691. PMID 18698067
- [Background] Kohrt BA, Kunz RD, Koirala NR. Validation of the Nepali version of beck anxiety inventory. Journal of Institute of Medicine. 2007 Jan 21;26(3).
- [Background] Linehan M. Cognitive-behavioral treatment of borderline personality disorder. Guilford press; 1993.
- [Background] Linehan MM. Skills training manual for treating borderline personality disorder. Guilford Press; 1993.
- [Background] Neacsiu AD, Rizvi SL, Vitaliano PP, Lynch TR, Linehan MM. The dialectical behavior therapy ways of coping checklist: development and psychometric properties. J Clin Psychol. 2010 Jun;66(6):563-82. doi: 10.1002/jclp.20685. PMID 20455249
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498